CLINICAL TRIAL: NCT01818596
Title: A Phase 3 Open-label Safety Study of Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Alafenamide Single-Tablet Regimen in HIV-1 Positive Patients With Mild to Moderate Renal Impairment
Brief Title: Open-label Safety Study of E/C/F/TAF (Genvoya®) in HIV-1 Positive Patients With Mild to Moderate Renal Impairment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-292-0112; 2013-000516-25 (EudraCT Number)
Record Dates: First submitted 2013-03-22; First posted 2013-03-26 (Estimated); Results first posted 2016-02-18 (Estimated); Last update posted 2020-03-02 (Actual); Status verified 2019-06

CONDITIONS: HIV; HIV Infections
Keywords: HIV; HIV-1 Infected; Treatment Experienced; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- E/C/F/TAF (Experimental): Participants will receive E/C/F/TAF for 144 weeks. Following Week 144, in countries where E/C/F/TAF is not available (except for the United Kingdom), participants will be given the option to continue in the study and receive E/C/F/TAF for another 48 weeks, or until the product becomes available through an access program, or until Gilead Sciences elects to discontinue the study in that country, whichever comes first.
  Interventions: Drug: E/C/F/TAF

INTERVENTIONS:
Drug: E/C/F/TAF — E/C/F/TAF (150/150/200/10 mg) FDC tablet administered orally once daily with food
  Other Names: Genvoya®

SUMMARY:
The primary objective of this study is to evaluate the effect of elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide (E/C/F/TAF) fixed-dose combination (FDC) tablet on renal parameters at Week 24 in treatment-naive and treatment-experienced HIV-positive, adults with mild to moderate renal impairment.

ELIGIBILITY:
Key Inclusion Criteria:

Cohort 1 (treatment-experienced switch)

* Must not have a history of known resistance to elvitegravir (EVG), tenofovir disoproxil fumarate (TDF), or emtricitabine (FTC)
* Plasma HIV-1 RNA concentrations (at least two measurements) at undetectable levels (according to the local assay being used) in the 6 months preceding the screening visit and have HIV-1 RNA < 50 copies/mL at screening
* Estimated glomerular filtration rate (GFR) 30-69 mL/min according to the Cockcroft-Gault formula for creatinine clearance, using actual weight
* May be currently enrolled in Gilead studies GS-US-236-0102, GS-US-236-0103, and GS-US-216-0114, but will be eligible to enroll only after the Week 144 visit for that study is complete; or currently receiving Stribild® (STB) or atazanavir (ATV)/cobicistat (COBI) + Truvada (TVD) in Gilead studies GS-US-236-0104 or GS-US-216-0105, but will be eligible to enroll only after the Week 48 visit for that study is complete.

Cohort 2 (treatment-naive)

* Plasma HIV-1 RNA levels ≥ 1,000 copies/mL at screening
* Screening genotype report provided by Gilead Sciences must show sensitivity to EVG, FTC, and TDF
* No prior use of any approved or investigational antiretroviral drug for any length of time, except the use for pre-exposure prophylaxis (PrEP), or post-exposure prophylaxis (PEP), up to 6 months prior to screening
* Estimated GFR 30-69 mL/min according to the Cockcroft Gault formula for creatinine clearance, using actual weight

All Cohorts:

All individuals must meet all of the following inclusion criteria to be eligible for participation in this study:

* The ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures
* CD4+ count of ≥ 50 cells/μL
* Stable renal function: serum creatinine measurements to be taken at least once (within three months of screening)
* Cause of underlying chronic kidney disease (eg hypertension, diabetes) stable, without change in medical management, for 3 months prior to baseline
* Normal electrocardiogram (ECG)
* Hepatic transaminases (AST and ALT) ≤ 5 x upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 mg/dL, or normal direct bilirubin
* Adequate hematologic function
* Serum amylase ≤ 5 x ULN
* Females of childbearing potential must agree to utilize highly effective contraception methods (two separate forms of contraception, one of which must be an effective barrier method, or be non-heterosexually active, practice sexual abstinence) from screening throughout the duration of study treatment and for 30 days following the last dose of study drug
* Females who utilize hormonal contraceptive as one of their birth control methods must have used the same method for at least three months prior to study dosing
* Males must agree to utilize a highly effective method of contraception during heterosexual intercourse throughout the study period and for 30 days following discontinuation of investigational medicinal product. A highly effective method of contraception is defined as two separate forms of contraception, one of which must be an effective barrier method, or males must be non-heterosexually active, or practice sexual abstinence

Key Exclusion Criteria:

* A new AIDS-defining condition (excluding CD4 cell count and percentage criteria) diagnosed within the 30 days prior to screening,with the exception of the first two bullet points
* Hepatitis C virus (HCV) antibody positive. Individuals who are HCV positive, but have a documented negative HCV RNA, are eligible
* Hepatitis B surface antigen (HBVsAg) positive
* Individuals receiving drug treatment for Hepatitis C, or individuals who are anticipated to receive treatment for Hepatitis C during the course of the study
* Individuals experiencing decompensated cirrhosis (eg, ascites, encephalopathy, etc.)
* Females who are breastfeeding
* Positive serum pregnancy test
* Have an implanted defibrillator or pacemaker
* Current alcohol or substance use judged by the Investigator to potentially interfere with study compliance
* A history of malignancy within the past 5 years or ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, non-invasive cutaneous squamous carcinoma
* Active, serious infections (other than HIV-1 infection) requiring parenteral antibiotic or antifungal therapy within 30 days prior to baseline
* Individuals on hemodialysis, other forms of renal replacement therapy, or on treatment for underlying kidney diseases (including prednisolone and dexamethasone)
* Individuals receiving ongoing therapy with any medications not to be used with EVG, COBI, FTC, or TAF or individuals with any known allergies to the excipients of E/C/F/TAF

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2013-03-27 (Actual); Primary Completion 2014-07-31 (Actual); Study Completion 2018-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (70):
- United States (51):
  - Maricopa Integrated Health System - McDowell Clinic, Phoenix, Arizona
  - Pueblo Family Physicians, Phoenix, Arizona
  - Health for Life Clinic PLLC, Little Rock, Arkansas
  - Pacific Oaks Medical Group, Beverly Hills, California
  - Kaiser Permanente, Hayward, California
  - Long Beach Education and Research Consultants, Long Beach, California
  - LA Gay & Lesbian Center - Jeffrey Goodman Special Care Clinic, Los Angeles, California
  - Peter J Ruane, MD, Inc, Los Angeles, California
  - Anthony Mills MD, Inc, Los Angeles, California
  - Desert Medical Group Inc. dba Desert Oasis Healthcare Medical Group, Palm Springs, California
  - Kaiser Permanente Medical Group, Sacramento, California
  - Metropolis Medical, San Francisco, California
  - Kaiser Permanente CTU San Francisco, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - National Jewish Health, Denver, Colorado
  - Dupont Circle Physician's Group, Washington D.C., District of Columbia
  - Gary J. Richmond, MD PA, Fort Lauderdale, Florida
  - Midway Immunology and Research Center, Ft. Pierce, Florida
  - Idocf/Valuhealthmd, Orlando, Florida
  - University of South Florida, Tampa, Florida
  - Triple O Research Institute, P.A., West Palm Beach, Florida
  - Rowan Tree Medical, P.A., Wilton Manors, Florida
  - Infectious Disease Specialists of Atlanta, Decatur, Georgia
  - Mercer University, Macon, Georgia
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Community Research Initiative of New England, Boston, Massachusetts
  - The Research Institute, Springfield, Massachusetts
  - Be Well Medical Center, P.C., Berkley, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - The Kansas City Care Clinic (KC Free Health Clinic), Kansas City, Missouri
  - Southampton Healthcare, Inc., St Louis, Missouri
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Saint Michael's Medical Center, Newark, New Jersey
  - Southwest CARE Center, Santa Fe, New Mexico
  - Albany Medical College, Albany, New York
  - Upstate Infectious Diseases Associates, Albany, New York
  - North Shore University Hospital/Division of Infectious Diseases, Manhasset, New York
  - Aids Care, Rochester, New York
  - Jacobi Medical Center, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of Cincinnati, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - University of PA HIV Clinical Trials Unit, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - St. Hope Foundation, Bellaire, Texas
  - North Texas Infectious Diseases Consultants, PA, Dallas, Texas
  - Garcias' Family Health Group, Harlingen, Texas
  - Therapeutic Concepts, PA, Houston, Texas
  - Gordon E. Crofoot MD, PA, Houston, Texas
  - Peter Shalit, MD, Seattle, Washington
- Australia (3):
  - Holdsworth House Medical Practice, Darlinghurst, New South Wales
  - Clinical Research Infectious Diseases Department- Alfred Hospital, Melbourne, Victoria
  - Prahran Market Clinic, Prahran, Victoria
- Instituto Dominicano de Estudios Virologicos (IDEV), Santo Domingo, Dominican Republic
- France (2):
  - Hopital de la Croix Rousse, Lyon
  - GHPS Service des maladies infectieuses et tropicales pavillon Laveran unité de recherche clinique, Paris
- Hospital Civil de Guadalajara Dr. Juan I. Menchaca, Guadalajara, Jalisco, Mexico
- University Medical Center Utrecht, Utrecht, Netherlands
- Spain (3):
  - Hospital Universitari de Bellvitge, Barcelona
  - Germans Trias i Pujol University Hospital, Barcelona
  - Hospital La Paz, Madrid
- Thailand (4):
  - HIV-NAT, Thai Red Cross AIDS Research Centre, Bangkok
  - Faculty of Medicine Ramathibodi Hospital, Mahidol University, Bangkok
  - Department of Preventive and Social Medicine, Faculty of Medicine, Siriraj Hospital, Bangkok
  - Srinagarind Hospital, Khon Kaen University, Khon Kaen
- United Kingdom (4):
  - Brighton & Sussex University Hospitals NHS Trust, Brighton
  - Kings College London, London
  - Chelsea and Westminster NHS Foundation Trust Hospital, London
  - Central Manchester University Hospitals NHS foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy

REFERENCES:
- [Result] Pozniak A, Arribas JR, Gathe J, Gupta SK, Post FA, Bloch M, Avihingsanon A, Crofoot G, Benson P, Lichtenstein K, Ramgopal M, Chetchotisakd P, Custodio JM, Abram ME, Wei X, Cheng A, McCallister S, SenGupta D, Fordyce MW; GS-US-292-0112 Study Team. Switching to Tenofovir Alafenamide, Coformulated With Elvitegravir, Cobicistat, and Emtricitabine, in HIV-Infected Patients With Renal Impairment: 48-Week Results From a Single-Arm, Multicenter, Open-Label Phase 3 Study. J Acquir Immune Defic Syndr. 2016 Apr 15;71(5):530-7. doi: 10.1097/QAI.0000000000000908. PMID 26627107
- [Result] Post FA, Tebas P, Clarke A, Cotte L, Short WR, Abram ME, Jiang S, Cheng A, Das M, Fordyce MW. Brief Report: Switching to Tenofovir Alafenamide, Coformulated With Elvitegravir, Cobicistat, and Emtricitabine, in HIV-Infected Adults With Renal Impairment: 96-Week Results From a Single-Arm, Multicenter, Open-Label Phase 3 Study. J Acquir Immune Defic Syndr. 2017 Feb 1;74(2):180-184. doi: 10.1097/QAI.0000000000001186. PMID 27673443

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in North America, Australia, Asia, and Europe. The first participant was screened on 27 March 2013. The last study visit occurred on 18 July 2018.
Pre-assignment Details: 380 participants were screened.
Groups:
- Cohort 1 (Treatment-experienced): Elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide (E/C/F/TAF) (150/150/200/10 mg) fixed-dose combination (FDC) tablet administered orally once daily with food for up to 240 weeks in antiretroviral treatment (ART)-experienced participants
- Cohort 2 (Treatment-naive): E/C/F/TAF (150/150/200/10 mg) FDC tablet administered orally once daily with food for up to 188 weeks in ART-naive participants
Period: Overall Study
Arm/Group | Cohort 1 (Treatment-experienced) | Cohort 2 (Treatment-naive)
Started | 246 | 6
Completed | 215 | 6
Not Completed | 31 | 0
Not completed — Enrolled but Not Treated | 4 | 0
Not completed — Adverse Event | 7 | 0
Not completed — Death | 3 | 0
Not completed — Investigator's Discretion | 4 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrew Consent | 5 | 0
Not completed — Lost to Follow-up | 7 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants were enrolled and received at least 1 dose of study drug
Groups:
- Cohort 1 (Treatment-experienced): E/C/F/TAF (150/150/200/10 mg) FDC tablet administered orally once daily with food for up to 240 weeks in ART-experienced participants
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (Treatment-experienced) | Cohort 2 (Treatment-naive) | Total
Number analyzed (Participants) | 242 | 6 | 248
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (9.9) | 55 (7.1) | 58 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 0 | 50
  Male | 192 | 6 | 198
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 34 | 1 | 35
  Race: American Indian or Alaska Native | 1 | 0 | 1
  Race: Black or African American | 44 | 3 | 47
  Race: Native Hawaiian or Pacific Islander | 2 | 0 | 2
  Race: White | 152 | 2 | 154
  Race: Other | 7 | 0 | 7
  Race: Not Permitted | 2 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 31 | 1 | 32
  Ethnicity: Not Hispanic or Latino | 209 | 5 | 214
  Ethnicity: Not Permitted | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 166 | 5 | 171
  United Kingdom | 5 | 0 | 5
  Thailand | 30 | 1 | 31
  Spain | 13 | 0 | 13
  Netherlands | 2 | 0 | 2
  Dominican Republic | 6 | 0 | 6
  Mexico | 2 | 0 | 2
  Australia | 12 | 0 | 12
  France | 6 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Estimated Glomerular Filtration Rate Calculated by the Cockcroft-Gault Formula (eGFR_CG) at Week 24
Description: eGFR is a measurement of the kidney's ability to filter blood.
Time Frame: Baseline; Week 24
Population: Participants in the Safety Analysis Set (enrolled and received at least 1 dose of study drug) with available data at the respective time point were analyzed.
Measure: Median (Inter-Quartile Range); unit: mL/min
Arm/Group | Cohort 1 (Treatment-experienced) | Cohort 2 (Treatment-naive)
Number analyzed (Participants) | 242 | 6
mL/min
  Baseline | 55.6 [45.7 to 62.4] | 60.2 [45.0 to 63.2]
  Change at Week 24: number analyzed (Participants) | 233 | 6
  Change at Week 24 | -0.4 [-4.7 to 4.5] | -0.3 [-3.6 to 1.3]

2. Primary Outcome: Change From Baseline in eGFR Calculated by the Chronic Kidney Disease Epidemiology Collaboration Method Based on Cystatin C (eGFR_CKD-EPI,cysC) at Week 24
Description: eGFR is a measurement of the kidney's ability to filter blood. The eGFR_CKD-EPI,cysC method is adjusted for age and sex.
Time Frame: Baseline; Week 24
Population: Participants in the Safety Analysis Set with available data at the respective time point were analyzed.
Measure: Median (Inter-Quartile Range); unit: mL/min/1.73 m^2
Arm/Group | Cohort 1 (Treatment-experienced) | Cohort 2 (Treatment-naive)
Number analyzed (Participants) | 242 | 6
mL/min/1.73 m^2
  Baseline: number analyzed (Participants) | 241 | 6
  Baseline | 69.7 [55.9 to 82.7] | 70.2 [64.0 to 100.8]
  Change at Week 24: number analyzed (Participants) | 231 | 6
  Change at Week 24 | 3.8 [-4.8 to 11.2] | 3.9 [-3.3 to 13.2]

3. Primary Outcome: Change From Baseline in eGFR Calculated by the CKD-EPI Method Based on Serum Creatinine (eGFR_CKD-EPI,Creatinine) at Week 24
Description: eGFR is a measurement of the kidney's ability to filter blood. The eGFR_CKD-EPI,creatinine method is adjusted for age, race, and sex.
Time Frame: Baseline; Week 24
Population: Participants in the Safety Analysis Set with available data at the respective time point were analyzed.
Measure: Median (Inter-Quartile Range); unit: mL/min/1.73 m^2
Arm/Group | Cohort 1 (Treatment-experienced) | Cohort 2 (Treatment-naive)
Number analyzed (Participants) | 242 | 6
mL/min/1.73 m^2
  Baseline | 54.1 [46.0 to 62.8] | 54.4 [41.7 to 81.4]
  Change at Week 24: number analyzed (Participants) | 233 | 6
  Change at Week 24 | -1.8 [-6.1 to 4.9] | -2.6 [-11.1 to -0.9]

4. Secondary Outcome: Change From Baseline in Actual GFR (aGFR) of E/C/F/TAF for Participants Enrolled in the PK/PD Substudy
Description: aGFR was directly measured using iohexol plasma clearance (CLiohexol).
Time Frame: Baseline; Week 2, 4, or 8; Week 24
Population: Participants in the Pharmacodynamic (PD) Substudy Analysis Set (enrolled in the pharmacokinetic (PK)/PD substudy, received at least 1 dose of study drug, and had baseline and at least 1 postbaseline assessment for aGFR assessed by CLiohexol) with available data at the respective time point were analyzed.
Measure: Mean (Standard Deviation); unit: mL/min
Groups:
- Substudy Participants: E/C/F/TAF (150/150/200/10 mg) FDC tablet administered orally once daily with food for up to 240 weeks
Arm/Group | Substudy Participants
Number analyzed (Participants) | 32
mL/min
  Baseline | 60.1 (19.06)
  Change at Week 2, 4, or 8 | -0.6 (8.45)
  Change at Week 24: number analyzed (Participants) | 30
  Change at Week 24 | 1.4 (9.91)
Statistical Analysis 1: Comparison: Substudy Participants; Comparison is made between the baseline value and the value from the Week 2, 4, or 8 visit and presented as a geometric least squares mean (GLSM) ratio with 90% confidence interval (CI). Postbaseline value and baseline value were used as test and reference, respectively; Test type: Non-Inferiority or Equivalence — 30 participants with evaluable aGFR (measured by iohexol clearance) in either cohort would provide at least 90% power to show that aGFR change is < 20% after participants were administered E/C/F/TAF. In this sample size/power computation, it was assumed that the intra-participant variation for aGFR is 0.17 mL/min on natural logarithm scale and a clinical meaningful boundary in aGFR change is 80% to 125%; Difference in GLSM Ratio = 98.94, 90% CI 2-sided [93.71 to 104.46] — A parametric analysis of variance model using a mixed-effects model with repeated statement was fitted to the natural logarithm transferred aGFR obtained at postbaseline visits and baseline
Statistical Analysis 2: Comparison: Substudy Participants; Comparison is made between the baseline value and the value from the Week 24 visit and presented as a GLSM ratio with 90% CI. Week 24 value and baseline value were used as test and reference, respectively; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Difference in GLSM Ratio = 102.66, 90% CI 2-sided [97.11 to 108.53] — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Percent Change From Baseline in C-type Collagen Sequence (CTX) at Weeks 24 and 48
Description: CTX is a biomarker of bone turnover.
Time Frame: Baseline; Weeks 24 and 48
Population: Participants in the Safety Analysis Set with available data at the respective time point were analyzed.
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | Cohort 1 (Treatment-experienced) | Cohort 2 (Treatment-naive)
Number analyzed (Participants) | 226 | 6
percentage change
  Change at Week 24 | -3.9 [-15.8 to 10.7] | 16.9 [0.0 to 21.7]
  Change at Week 48: number analyzed (Participants) | 222 | 6
  Change at Week 48 | -2.2 [-16.7 to 24.4] | 0.0 [-4.8 to 10.8]

6. Secondary Outcome: Percent Change From Baseline in Procollagen Type 1 N-terminal Propeptide (P1NP) at Weeks 24 and 48
Description: P1NP is a biomarker of bone turnover.
Time Frame: Baseline; Weeks 24 and 48
Population: Participants in the Safety Analysis Set with available data at the respective time point were analyzed.
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | Cohort 1 (Treatment-experienced) | Cohort 2 (Treatment-naive)
Number analyzed (Participants) | 229 | 6
percentage change
  Change at Week 24 | -12.98 [-34.48 to 8.86] | 6.44 [-5.08 to 47.62]
  Change at Week 48: number analyzed (Participants) | 224 | 6
  Change at Week 48 | -25.29 [-45.98 to 2.00] | 2.27 [-29.12 to 41.80]

7. Secondary Outcome: Percent Change From Baseline in Retinol Binding Protein (RBP) to Creatinine Ratio (μg/g) at Weeks 24, 48, 96, and 144
Description: Urine RBP is a renal biomarker which is used to evaluate drug-induced kidney injury.
Time Frame: Baseline; Weeks 24, 48, 96, and 144
Population: Participants in the Safety Analysis Set with available data at the respective time point were analyzed.
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | Cohort 1 (Treatment-experienced) | Cohort 2 (Treatment-naive)
Number analyzed (Participants) | 227 | 6
percentage change
  Change at Week 24 | -56.2 [-90.0 to -11.8] | 68.8 [-37.1 to 72.6]
  Change at Week 48: number analyzed (Participants) | 220 | 6
  Change at Week 48 | -68.9 [-92.2 to -20.5] | 47.8 [13.3 to 78.9]
  Change at Week 96: number analyzed (Participants) | 212 | 6
  Change at Week 96 | -64.1 [-91.4 to 9.8] | 55.0 [-10.5 to 197.0]
  Change at Week 144: number analyzed (Participants) | 187 | 6
  Change at Week 144 | -63.8 [-92.4 to 4.6] | -1.0 [-10.2 to 43.4]

8. Secondary Outcome: Percent Change From Baseline in Urine Beta-2-microglobulin to Creatinine Ratio (μg/g) at Weeks 24, 48, 96, and 144
Description: Urine beta-2-microglobulin is a renal biomarker which is used to evaluate drug-induced kidney injury.
Time Frame: Baseline; Weeks 24, 48, 96, and 144
Population: Participants in the Safety Analysis Set with available data at the respective time point were analyzed.
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | Cohort 1 (Treatment-experienced) | Cohort 2 (Treatment-naive)
Number analyzed (Participants) | 224 | 6
percentage change
  Change at Week 24 | -70.7 [-92.6 to -11.1] | -19.5 [-93.0 to 81.3]
  Change at Week 48: number analyzed (Participants) | 214 | 6
  Change at Week 48 | -76.5 [-94.6 to -17.7] | -59.2 [-85.0 to 34.3]
  Change at Week 96: number analyzed (Participants) | 210 | 6
  Change at Week 96 | -83.6 [-96.4 to -31.1] | -45.9 [-95.8 to 195.6]
  Change at Week 144: number analyzed (Participants) | 185 | 6
  Change at Week 144 | -81.9 [-95.5 to -18.0] | -3.6 [-66.7 to 73.5]

9. Secondary Outcome: Percentage of Participants Experiencing Adverse Events or Graded Laboratory Abnormalities
Description: Adverse events (AEs) and graded laboratory abnormalities occurring during the E/C/F/TAF treatment period were summarized across the participant population. A participant was counted once if they had a qualifying event.
Time Frame: Baseline up to Week 240 plus 30 days
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 (Treatment-experienced) | Cohort 2 (Treatment-naive)
Number analyzed (Participants) | 242 | 6
percentage of participants
  Any AE | 95.5 | 100.0
  Grade 3 or 4 AE | 22.3 | 16.7
  AE leading to drug discontinuation | 5.0 | 0
  Serious AE | 22.7 | 16.7
  Grade 3 or 4 laboratory abnormality | 42.6 | 66.7

10. Secondary Outcome: Percentage of Participants Achieving HIV-1 RNA < 50 Copies/mL at Weeks 24, 48, 96, and 144
Description: The percentage of participants achieving HIV-1 RNA < 50 Copies/mL at Weeks 24, 48, 96, and 144 was analyzed using the snapshot algorithm, which defines a patient's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Weeks 24, 48, 96, and 144
Population: Full Analysis Set included participants who were enrolled and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 (Treatment-experienced) | Cohort 2 (Treatment-naive)
Number analyzed (Participants) | 242 | 6
percentage of participants
  Week 24 | 95.0 | 83.3
  Week 48 | 93.0 | 100.0
  Week 96 | 88.4 | 100.0
  Week 144 | 81.4 | 100.0

11. Secondary Outcome: Pharmacokinetic (PK) Parameter: Cmax of TAF
Description: Cmax is defined as the maximum concentration of drug. Blood draws for this outcome may have been at the Week 2, 4, or 8 visit.
Time Frame: Predose, and 5 minutes, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 8, and 24 hours postdose
Population: Participants in the PK Substudy Analysis Set (enrolled in the PK/PD substudy, received at least 1 dose of study drug, and for whom steady-state PK parameters were available) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Substudy Participants
Number analyzed (Participants) | 30
ng/mL | 269.8 (180.77)

12. Secondary Outcome: PK Parameter: Tmax of TAF
Description: Tmax is defined as the time of Cmax. Blood draws for this outcome may have been at the Week 2, 4, or 8 visit.
Time Frame: Predose, and 5 minutes, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 8, and 24 hours postdose
Population: Participants in the PK Substudy Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Substudy Participants
Number analyzed (Participants) | 30
hours | 0.97 [0.50 to 1.98]

13. Secondary Outcome: PK Parameter: Clast of TAF
Description: Clast is defined as the last observable concentration of drug. Blood draws for this outcome may have been at the Week 2, 4, or 8 visit.
Time Frame: Predose, and 5 minutes, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 8, and 24 hours postdose
Population: Participants in the PK Substudy Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Substudy Participants
Number analyzed (Participants) | 30
ng/mL | 7.6 (25.73)

14. Secondary Outcome: PK Parameter: Tlast of TAF
Description: Tlast is defined as the time of Clast. Blood draws for this outcome may have been at the Week 2, 4, or 8 visit.
Time Frame: Predose, and 5 minutes, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 8, and 24 hours postdose
Population: Participants in the PK Substudy Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Substudy Participants
Number analyzed (Participants) | 30
hours | 4.45 [3.82 to 5.00]

15. Secondary Outcome: PK Parameter: λz of TAF
Description: λz is defined as the terminal elimination rate constant. Blood draws for this outcome may have been at the Week 2, 4, or 8 visit.
Time Frame: Predose, and 5 minutes, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 8, and 24 hours postdose
Population: Participants in the PK Substudy Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | Substudy Participants
Number analyzed (Participants) | 30
1/hour | 1.764 (1.4521)

16. Secondary Outcome: PK Parameter: AUCtau of TAF
Description: AUCtau is defined as the concentration of drug over time (area under the plasma concentration versus time curve over the dosing interval). Blood draws for this outcome may have been at the Week 2, 4, or 8 visit.
Time Frame: Predose, and 5 minutes, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 8, and 24 hours postdose
Population: Participants in the PK Substudy Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Substudy Participants
Number analyzed (Participants) | 30
ng*h/mL | 368.4 (631.20)

17. Secondary Outcome: PK Parameter: t1/2 of TAF
Description: t1/2 is defined as the estimate of the terminal elimination half-life of the drug. Blood draws for this outcome may have been at the Week 2, 4, or 8 visit.
Time Frame: Predose, and 5 minutes, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 8, and 24 hours postdose
Population: Participants in the PK Substudy Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Substudy Participants
Number analyzed (Participants) | 30
hours | 0.43 [0.37 to 0.52]

18. Secondary Outcome: PK Parameter: AUCtau of Tenofovir Diphosphate (TFV-DP) in Peripheral Blood Mononuclear Cell (PBMC) for Participants Enrolled in PK/PD Sub-study
Description: TFV-DP is an active phosphorylated metabolite of tenofovir alafenamide. AUCtau is defined as the concentration of drug over time (area under the plasma concentration versus time curve over the dosing interval). Blood draws for this outcome may have been at the Week 2, 4, or 8 visit.
Time Frame: Predose, and 5 minutes, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 8, and 24 hours postdose
Population: Participants who were enrolled in the PK/PD substudy, received at least 1 dose of study drug, and for whom the steady-state PK parameter (AUCtau) of TFV-DP was evaluable were analyzed.
Measure: Mean (Standard Deviation); unit: µmol*h/L
Arm/Group | Substudy Participants
Number analyzed (Participants) | 23
µmol*h/L | 50.6 (55.75)

19. Secondary Outcome: Change From Baseline in the eGFR_CG at Weeks 48, 96, and 144
Description: eGFR is a measurement of the kidney's ability to filter blood.
Time Frame: Baseline; Weeks 48, 96, and 144
Population: Participants in the Safety Analysis Set with available data at the respective time point were analyzed.
Measure: Median (Inter-Quartile Range); unit: mL/min
Arm/Group | Cohort 1 (Treatment-experienced) | Cohort 2 (Treatment-naive)
Number analyzed (Participants) | 242 | 6
mL/min
  Baseline | 55.6 [45.7 to 62.4] | 60.2 [45.0 to 63.2]
  Change at Week 48: number analyzed (Participants) | 225 | 5
  Change at Week 48 | -0.6 [-5.4 to 5.4] | -0.6 [-1.9 to 4.2]
  Change at Week 96: number analyzed (Participants) | 217 | 6
  Change at Week 96 | 0.6 [-4.6 to 7.2] | -1.9 [-4.0 to 6.0]
  Change at Week 144: number analyzed (Participants) | 206 | 6
  Change at Week 144 | 1.5 [-4.8 to 7.2] | 7.0 [3.3 to 11.2]

20. Secondary Outcome: Change From Baseline in eGFR_CKD-EPI,cysC at Weeks 48, 96, and 144
Description: eGFR is a measurement of the kidney's ability to filter blood. The eGFR_CKD-EPI,cysC method is adjusted for age and sex.
Time Frame: Baseline; Weeks 48, 96, and 144
Population: Participants in the Safety Analysis Set with available data at the respective time point were analyzed.
Measure: Median (Inter-Quartile Range); unit: mL/min/1.73 m^2
Arm/Group | Cohort 1 (Treatment-experienced) | Cohort 2 (Treatment-naive)
Number analyzed (Participants) | 242 | 6
mL/min/1.73 m^2
  Baseline: number analyzed (Participants) | 241 | 6
  Baseline | 69.7 [55.9 to 82.7] | 70.2 [64.0 to 100.8]
  Change at Week 48: number analyzed (Participants) | 224 | 5
  Change at Week 48 | 1.7 [-7.3 to 12.0] | 7.3 [-0.1 to 12.2]
  Change at Week 96: number analyzed (Participants) | 216 | 6
  Change at Week 96 | 3.2 [-3.6 to 11.8] | 5.6 [-7.2 to 20.8]
  Change at Week 144: number analyzed (Participants) | 205 | 6
  Change at Week 144 | 3.1 [-4.8 to 11.8] | 3.5 [-1.8 to 22.9]

21. Secondary Outcome: Change From Baseline in eGFR_CKD-EPI,Creatinine at Weeks 48, 96, and 144
Description: as for outcome 3
Time Frame: Baseline; Weeks 48, 96, and 144
Population: Participants in the Safety Analysis Set with available data at the respective time point were analyzed.
Measure: Median (Inter-Quartile Range); unit: mL/min/1.73 m^2
Arm/Group | Cohort 1 (Treatment-experienced) | Cohort 2 (Treatment-naive)
Number analyzed (Participants) | 242 | 6
mL/min/1.73 m^2
  Baseline | 54.1 [46.0 to 62.8] | 54.4 [41.7 to 81.4]
  Change at Week 48: number analyzed (Participants) | 226 | 5
  Change at Week 48 | -1.7 [-7.9 to 4.2] | -3.0 [-4.9 to 0.6]
  Change at Week 96: number analyzed (Participants) | 217 | 6
  Change at Week 96 | 0.1 [-5.7 to 6.4] | -3.1 [-9.5 to 2.1]
  Change at Week 144: number analyzed (Participants) | 206 | 6
  Change at Week 144 | 1.7 [-5.3 to 8.5] | 0.9 [-5.7 to 6.0]

ADVERSE EVENTS:
Time Frame: First dose date up to Week 240 plus 30 days
Description: Safety Analysis Set included participants were enrolled and received at least 1 dose of study drug.
Arm/Group | Cohort 1 (Treatment-experienced) | Cohort 2 (Treatment-naive)
Serious Adverse Events (participants affected / at risk) | 55/242 | 1/6
Other Adverse Events (participants affected / at risk) | 195/242 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (Treatment-experienced) (N=242) | Cohort 2 (Treatment-naive) (N=6)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 4 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0
Blindness unilateral (Eye disorders) | 1 | 0
Vitreous detachment (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Abscess neck (Infections and infestations) | 1 | 0
Acute hepatitis c (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 2 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Endophthalmitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 0
Gastrointestinal viral infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 1 | 0
Ophthalmic herpes zoster (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervical radiculopathy (Nervous system disorders) | 1 | 0
Facial paralysis (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Drug dependence (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (Treatment-experienced) (N=242) | Cohort 2 (Treatment-naive) (N=6)
Supraventricular extrasystoles (Cardiac disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 16 | 0
Diarrhoea (Gastrointestinal disorders) | 32 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 22 | 0
Vomiting (Gastrointestinal disorders) | 13 | 0
Chest pain (General disorders) | 10 | 1
Fatigue (General disorders) | 20 | 1
Peripheral swelling (General disorders) | 8 | 1
Bronchitis (Infections and infestations) | 37 | 1
Hordeolum (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 10 | 1
Nasopharyngitis (Infections and infestations) | 25 | 0
Sinusitis (Infections and infestations) | 18 | 0
Upper respiratory tract infection (Infections and infestations) | 39 | 1
Urinary tract infection (Infections and infestations) | 25 | 0
Exposure to communicable disease (Injury, poisoning and procedural complications) | 1 | 1
Cardiac murmur (Investigations) | 1 | 1
Electrocardiogram st-t change (Investigations) | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 5 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 7 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1
Vitamin d deficiency (Metabolism and nutrition disorders) | 4 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 34 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 27 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 26 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 13 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 25 | 2
Tendonitis (Musculoskeletal and connective tissue disorders) | 5 | 1
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Dizziness (Nervous system disorders) | 18 | 0
Headache (Nervous system disorders) | 20 | 1
Migraine (Nervous system disorders) | 2 | 1
Paraesthesia (Nervous system disorders) | 13 | 0
Somnolence (Nervous system disorders) | 3 | 1
Proteinuria (Renal and urinary disorders) | 3 | 1
Renal cyst (Renal and urinary disorders) | 14 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 6 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 24 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 4 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 1
Rash (Skin and subcutaneous tissue disorders) | 15 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 1
Hypertension (Vascular disorders) | 24 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 1

LIMITATIONS AND CAVEATS:
Enrollment in Cohort 2 (treatment-naive) was low, which affects the interpretation of the data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years